CLINICAL TRIAL: NCT00469573
Title: Safety and Efficacy of Optive in Contact Lens Wearers With Dry Eyes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Jodi Luchs, MD, South Shore Eye Care
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 5302
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

ARMS (1):
- 1. (Other)
  Interventions: Drug: 1. Optive

INTERVENTIONS:
Drug: 1. Optive — Optive 15ml- (in the eye) Instill one drop twice daily in each eye

SUMMARY:
The purpose of this study is to determine if Optive®eye drops are safe for people who wear contact lenses and have dry eyes. The second goal of the study is to determine if using Optive®eye drops can improve my dry eye scores on a standard dry eye test (called the OSDI).

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 and over

  * Self-reported use of daily-wear soft contact lenses that have been a proper fit for at least one month prior to the screening visit.
  * Complaint of dry eyes
  * OSDI score > 23

Exclusion Criteria:

* Use of RGP or PMMA contact lenses

  * Poorly fitting contact lenses
  * Concurrent ocular conditions or pathology that could affect contact lens fit or patient's ability to complete study
  * Concurrent use of topical medications other than study medications
  * Use of systemic medications with ocular drying sequelae:

    * Antihistamines
    * Decongestants
    * Antispasmotics Antidepressants Change in contact lens care solutions within the prior 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety | 8 months

SECONDARY OUTCOMES:
Efficacy | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Luchs, MD, Principal Investigator — South Shore Eye Care
Locations (1):
- South Shore Eye Care, Wantagh, New York, United States